CLINICAL TRIAL: NCT01278212
Title: A Phase II Study of Accelerated Hypofractionated Radiotherapy (AHF-RT) After Breast Conserving Surgery (BCS) in Medically Underserved Patients
Brief Title: Accelerated Hypofractionated Radiotherapy (AHF-RT) for the Treatment of Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Principal Investigator, Harriet Eldredge-Hindy, Assistant Professor, M.D., University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10.0584; BCC-AHF-RT-10 (Other: James Graham Brown Cancer Center Clinical Trials Office)
Record Dates: First submitted 2011-01-12; First posted 2011-01-17 (Estimated); Results first posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; breast neoplasm; breast tumor; radiotherapy; radiation; accelerated; lumpectomy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AHF-RT (Experimental): accelerated hypofractionated radiotherapy (AHF-RT)
  30 Gy in 5 fractions once a week for 5 weeks, followed by optional boost of 10-16 Gy
  Interventions: Radiation: accelerated hypofractionated radiotherapy (AHF-RT)

INTERVENTIONS:
Radiation: accelerated hypofractionated radiotherapy (AHF-RT) — 30 Gy in 5 fractions once a week for 5 weeks, followed by optional boost of 10-16 Gy
  Other Names: accelerated hypofractionated radiation

SUMMARY:
The goal of this study is to explore the safety, effectiveness, quality of life, and cost effectiveness of accelerated hypofractionated radiotherapy (AHF-RT) as treatment after lumpectomy in patients with early stage breast cancer.

DETAILED DESCRIPTION:
The traditional radiation treatment schedule for patients who have had a lumpectomy for early stage breast cancer is 15 to 30 treatments delivered once a day for 3 to 6 weeks. This treatment schedule can be inconvenient and costly for elderly, rural, uninsured, and minority patients. This study will evaluate a new radiation treatment schedule called whole-breast accelerated hypofractionated radiotherapy (AHF-RT). AHF-RT delivers higher doses of radiation in fewer treatments than traditional radiation therapy. The AHF-RT treatment course is completed with 5 radiation treatments delivered once a week for 5 weeks.

The purpose of this study is to determine if accelerated hypofractionated radiotherapy (AHF-RT) is a safe, effective, more convenient, and less costly alternative to traditional radiation that will offer the same chance of cure with no additional side effects.

ELIGIBILITY:
Inclusion Criteria:

Only women who satisfy all of the following conditions will be eligible for this study.

1. must consent to be in the study and must have signed an approved consent form conforming with federal and institutional guidelines
2. must be at least 21 years old
3. must have stage 0, I, or II breast cancer
4. On histological examination, the tumor must be ductal carcinoma in situ (DCIS) or invasive adenocarcinoma of the breast.
5. Surgical treatment of the breast must have been breast conserving surgery (BCS). The margins of the resected specimen must be histologically free of tumor (including DCIS component). Reexcision of surgical margins is permitted.
6. Gross disease may be unifocal or multifocal with pathologic (invasive and/or DCIS) tumor size excised with negative margins.
7. Patients with invasive breast cancer are required to have axillary staging which can include sentinel node biopsy alone (if sentinel node is negative), sentinel node biopsy followed by axillary dissection or sampling with a minimum total of 6 axillary nodes (if sentinel node is positive), or axillary dissection alone (with a minimum of 6 axillary nodes). Axillary staging is not required for patients with DCIS.
8. must begin adjuvant therapy (chemotherapy or radiotherapy) within 9 weeks following the last surgery for breast cancer (lumpectomy, re-excision of margins, or axillary staging procedure)
9. Patients must have all usual and customary hormone receptor (ER/PR) and estrogen receptor (ER) analysis performed on the primary tumor prior to enrollment. Patients with invasive disease must have HER2 receptor status determined (positive or negative) with immuno-histochemistry (IHC) and/or fluorescent in-situ hybridization (FISH).
10. At the time of study enrollment, patients must have had a history & physical exam within 4 months and a bilateral mammogram within 6 months.
11. Patients with a history of non-breast malignancies are eligible if they have been disease-free for 5 or more years prior to enrollment and are deemed by their physician to be at low risk for recurrence. Patients with the following cancers are eligible if diagnosed and treated within the past 5 years: carcinoma in situ of the cervix, carcinoma in situ of the colon, melanoma in situ, and basal cell and squamous cell carcinoma of the skin.
12. Patients must live in a county that is designated as Appalachian and/or rural by Kentucky Cancer Registry Criteria (see list below) and/or must hold their primary residence at least 10 miles from the nearest radiation facility. Patients who do not fit these criteria may still be considered eligible if they are determined to suffer significant financial and/or transportation hardship during a typical course of CF-RT or HF-RT (in the judgment of any of their treating physicians). Patients who live outside the Commonwealth of Kentucky are eligible if they fit any of these aforementioned conditions.

    * Appalachian counties in KY include: Adair, Bath, Bell, Boyd, Breathitt, Carter, Casey, Clark, Clay, Clinton, Cumberland, Edmonson, Elliott, Estill, Fleming, Floyd, Garrard, Green, Greenup, Harlan, Hart, Jackson, Johnson, Knott, Knox, Laurel, Lawrence, Lee, Leslie, Letcher, Lewis, Lincoln, Madison, Magoffin, Martin, McCreary, Menifee, Metcalfe, Monroe, Montgomery, Morgan, Nicholas, Owsley, Perry, Pike, Powell, Pulaski, Robertson, Rockcastle, Rowan, Russell, Wayne, Whitley, Wolfe.

Exclusion Criteria:

Men are not eligible for this study. Women with one or more of the following conditions are ineligible for this study.

1. T3, stage III, or stage IV breast cancer
2. More than 3 histologically positive axillary nodes
3. Axillary nodes with definite evidence of microscopic or macroscopic extracapsular extension
4. One or more positive non-axillary sentinel node(s) (Note that intramammary nodes are staged as axillary nodes.)
5. Palpable or radiographically suspicious ipsilateral or contralateral axillary, supraclavicular, infraclavicular, or internal mammary nodes, unless there is histologic confirmation that these nodes are negative for tumor
6. Suspicious microcalcifications, densities, or palpable abnormalities (in the ipsilateral or contralateral breast) unless biopsied and found to be benign
7. Non-epithelial breast malignancies such as sarcoma or lymphoma
8. Proven multicentric carcinoma (invasive cancer or DCIS) in more than one quadrant or separated by 4 or more centimeters
9. Paget's disease of the nipple
10. Synchronous bilateral invasive or non-invasive breast cancer
11. History of invasive breast cancer or DCIS (Patients with a history of lobular carcinoma in situ (LCIS) treated by surgery alone are eligible.)
12. Surgical margins that cannot be microscopically assessed or are positive at pathologic evaluation (If surgical margins are rendered free of disease by reexcision, the patient is eligible.)
13. Treatment plan that includes regional nodal irradiation
14. Current therapy with any hormonal agents such as raloxifene (Evista®), tamoxifen, or other selective estrogen receptor modulators (SERMs), either for osteoporosis or breast cancer prevention (Patients are eligible only if these medications are discontinued prior to enrollment.)
15. Cosmetic breast implants (Patients who have had implants removed are eligible.)
16. Prior breast or thoracic RT for any condition
17. Collagen vascular disease, specifically dermatomyositis with a CPK level above normal or with an active skin rash, systemic lupus erythematosis, or scleroderma
18. Pregnancy or lactation at the time of proposed randomization. Women of reproductive potential must agree to use an effective non-hormonal method of contraception during therapy.
19. Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2011-01; Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harriet Eldredge-Hindy, MD, Principal Investigator — James Graham Brown Cancer Center
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment 2011-2016, recruitment now complete
Groups:
- AHF-RT With Chemotherapy: If chemotherapy indicated: accelerated hypofractionated radiotherapy (AHF-RT)
  30 Gy in 5 fractions once a week for 5 weeks, followed by optional boost of 10-16 Gy
  accelerated hypofractionated radiotherapy (AHF-RT): 30 Gy in 5 fractions once a week for 5 weeks, followed by optional boost of 10-16 Gy
Period: Overall Study
Arm/Group | AHF-RT With Chemotherapy
Started | 158 (2011)
Completed | 158 (November 2020)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- AHF-RT: accelerated hypofractionated radiotherapy (AHF-RT)
  30 Gy in 5 fractions once a week for 5 weeks, followed by optional boost of 10-16 Gy
  accelerated hypofractionated radiotherapy (AHF-RT): 30 Gy in 5 fractions once a week for 5 weeks, followed by optional boost of 10-16 Gy
Arm/Group | AHF-RT
Number analyzed (Participants) | 158
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 100
  >=65 years | 58
Age, Continuous [Mean (Full Range); unit: years] | 59 [30 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 34
  White | 124
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 158
Tumor Subtypes [Count of Participants; unit: Participants] — invasive ductal carcinoma, invasive lobular carcinoma, ductal carcinoma in situ, and other less common types of carcinoma.
  Participants
    invasive ductal carcinoma | 102
    invasive lobular carcinoma | 16
    ductal carcinoma in situ | 35
    other less common types of carcinoma | 5
tumor grade [Count of Participants; unit: Participants] — Tumor grade was I, II, or III and was determined from surgical pathology from the time of lumpectomy. Grade 3 is worst outcome.
  Participants
    Grade 1 | 33
    Grade 2 | 67
    Grade 3 worst outcome | 58
stage [Count of Participants; unit: Participants] — Stage was 0, IA, IB, IIA, IIB, or III and was based on AJCC 7th edition staging manual. The higher the stage the worse the outcome.
  Participants
    Stage 0 | 36
    stage 1 | 89
    stage 2 | 33
    stage 3 | 0
Estrogen receptor status [Count of Participants; unit: Participants]
  + Estrogen receptor | 130
  - Estrogen receptor | 28

OUTCOME MEASURES:

1. Primary Outcome: Ipsilateral Breast Tumor Recurrence (IBTR)
Description: Both invasive and non-invasive IBTRs will be considered in calculating the primary endpoint.
Time Frame: at 5 years post completion of AHF-RT
Measure: Number; unit: percentage of participants
Arm/Group | AHF-RT
Number analyzed (Participants) | 158
percentage of participants | 2.7

ADVERSE EVENTS:
Time Frame: median follow up 5.5 years, (range, 0.2-9.9 years)
Description: Common Terminology Criteria for Adverse Events version 3.0
Arm/Group | AHF-RT
All-Cause Mortality (participants affected / at risk) | 17/158
Serious Adverse Events (participants affected / at risk) | 20/158
Other Adverse Events (participants affected / at risk) | 0/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AHF-RT (N=158)
Breast shrinkage or fibrosis (Reproductive system and breast disorders) | 17
cardiomyopathy (Cardiac disorders) | 1
Breast pain (Reproductive system and breast disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-12-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT01278212/Prot_SAP_000.pdf